CLINICAL TRIAL: NCT06363201
Title: Exploratory Study to Evaluate the Effect and Safety of the Use of Ocoxin Oral Solution on the Quality of Life of Paediatric Patients With Advanced Stage Solid Tumours
Brief Title: Effect and Safety of Ocoxin Oral Solution on the Quality of Life of Paediatric Patients With Advanced Stage Solid Tumours
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAT2024/PED01
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Advanced Cancer; Advanced Solid Tumor; Lymphoma, Hodgkin; Central Nervous System Tumor; Sarcoma; Germ Cell Tumor; Pediatric Cancer
Keywords: Epigallocatechin gallate; Paediatric; Advanced Solid Tumor; Quality of Life
MeSH Terms: conditions — Hodgkin Disease; Central Nervous System Neoplasms; Sarcoma; Neoplasms, Germ Cell and Embryonal; Neoplasms | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocoxin Oral Solution (Experimental): Patients will receive one vial of Ocoxin® daily from the start of oncospecific therapy until two weeks after the end of therapy.
  Interventions: Dietary Supplement: Ocoxin Oral solution

INTERVENTIONS:
Dietary Supplement: Ocoxin Oral solution — Patients will receive one vial of Ocoxin® orally daily, preferably at the same time each day. The duration of treatment will depend on the chemotherapy schedule the patient will receive. Treatment with Ocoxin® will be from the start of oncospecific therapy until two weeks after the end of therapy.

SUMMARY:
Exploratory study to evaluate the effect and safety of the use of Ocoxin® oral solution on the quality of life of paediatric patients with advanced stage solid tumours.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-centre, exploratory study in paediatric patients with advanced stage solid tumours receiving oncospecific therapy.

Ocoxin®: The research product, registered as a nutritional supplement (Ocoxin®, oral solution), manufactured by Catalysis S.L. of Spain. It comes in the form of 30 ml single-dose vials.

Forty paediatric patients will be included, distributed as follows: Hodgkin's lymphoma (10), Central Nervous System tumours (10), Sarcoma of any type (10) or Germinal Tumours (10).

Patients will receive one vial of Ocoxin® daily from the start of oncospecific therapy until two weeks after the end of therapy.

Prior to the start of treatment and before each cycle of QT, a haemogram and haemochemistry including albumin, total proteins, transaminases (TGO, TGP) will be performed. Physical examinations will be performed, and the patient's vital signs and body weight will be evaluated.

Prior to the start of treatment, in month three and four weeks after the end of oncospecific therapy, a CT scan will be performed (depending on the type of tumour, the system for evaluating the efficacy of the oncospecific treatment will be adapted).

Quality of life will be assessed using the paediatric quality of life questionnaire (PedsQLTm, version 4.0. Spanish). The questionnaire will be administered to the parent or guardian prior to the start of treatment, at month 3 and at the end of treatment with Ocoxin®. In the case of longer treatment regimens, intermediate quality of life measurements may be taken after the three months and before the end of treatment.

The influence of Ocoxin® Oral solution on the prevention of admissions due to toxicity attributable to cancer-specific therapy and changes in the patient's nutritional status will also be assessed.

Safety will be assessed by collecting adverse events (AEs), analytical parameters, physical examinations and vital signs.

Effect and safety variables will be summarised using descriptive statistics and frequency counts.

ELIGIBILITY:
Inclusion Criteria:

* Patient of either sex in the paediatric age group, between 7 and 18 years of age.
* Father, mother or legal guardian who consents in writing to the minor's participation in the study. Written consent of the minor for ages 12 to 18 years. Verbal consent of the minor for ages 7 to 11 years.
* Histologically confirmed diagnosis of solid tumour of any location, in advanced stage, with criteria to receive oncospecific therapy.
* Patients with haematological parameters within normal figures that allow them to receive oncospecific therapy, according to the management protocols for each of the diseases.

Exclusion Criteria:

* Pregnancy or breast-feeding (if less than 3 months have elapsed since delivery, abortion, or breast-feeding prior to the start of treatment).
* Hypersensitivity to any component of the product under study (Ocoxin®).
* Any disease or condition that could interfere with the interpretation of the results.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-28 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | 7 months
  Qualitative and quantitative data collection. To assess the effect of Ocoxin® on the quality of life of paediatric patients with advanced solid tumours by the Paediatric Quality of Life Questionnaire (PedsQLTm, version 4.0. Spanish). The questionnaire will be administered to the parent or guardian prior to the start of treatment, at month 3 and at the end of treatment with Ocoxin®. In the case of longer treatment regimens, intermediate quality of life measurements may be taken after the three-month treatment and before the end of treatment.

SECONDARY OUTCOMES:
Degree of toxicity related to oncospecific treatment | 7 months
  Qualitative and quantitative data collection. To evaluate the influence of Ocoxin® in the prevention of admissions due to toxicity to cancer-specific therapy (NCI-CTC scales). Admissions for toxicity. Information related to the need for admissions for mucositis (World Health Organization mucositis grade) or other causes shall be collected at each assessment during treatment and at the final assessment.
Nutritional Status | 7 months
  Qualitative and quantitative data collection. Changes in nutritional status. This will be assessed through body mass index (BMI) behavior at baseline, intermediate assessments, and final assessments.
Presence of Adverse Events (AE) | 7 months
  Qualitative and quantitative data collection. Product and non-product related adverse events described and classified as follows:
  Occurrence of any AE: yes/no Type: described according to the CTC nomenclature version 5.0 Duration: To be assessed by the start and end dates of the adverse event Intensity: To be assessed by the categories mild, moderate, severe, serious life-threatening or disabling, or serious life-threatening.
  Causality: assessed as highly probable/certain, probable, possible, possible, unlikely, unrelated, and not assessable/unclassifiable Severity: yes/no. In case of yes, it will be classified according to the categories of: causes death of the patient, threatens life, requires hospitalisation or prolongs an existing hospitalisation, causes disability, significant or persistent disability, causes a birth defect or congenital anomaly.
  Outcome: To be assessed according to the categories of recovered, improved, persists or sequelae.
Metabolic Status | 7 months
  Qualitative and quantitative data collection. The metabolic status of patients will be assessed by laboratory tests. The tests described in the evaluations will be performed according to the study schedule (haemogram, albumin, total proteins, TGP, TGO). They will be classified as normal, non-clinically significant abnormal and clinically significant abnormal. Clinically significant abnormal findings in laboratory parameters will be reported as AE.
Physical Status | 7 months
  Qualitative data collection. The physical status of patients shall be assessed by physical examination. The patient will be examined prior to study initiation, at on-treatment assessments, and at the end-of-treatment assessment. Any positive findings of clinical relevance on physical examination will be considered as an adverse event and will be described and classified as defined in the protocol for this type of event.
Response to oncospecific treatment | 7 months
  Qualitative data collection (the evaluation method used will also include RECIST criteria, iRECIST criteria, Cheeson criteria or other, in which case the method will be specified). Objective response to oncospecific treatment will be assessed by characterising the type of response after clinical evaluation of the patient at the end of the chemotherapy regimen. This will be classified as complete response, partial response, disease stabilisation or progression, following the response criteria established for each treatment protocol according to the underlying disease treated.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Escuela, Tegucigalpa (Honduras), Tegucigalpa, Francisco Morazán Department, Honduras

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Steliarova-Foucher E, Colombet M, Ries LAG, Moreno F, Dolya A, Bray F, Hesseling P, Shin HY, Stiller CA; IICC-3 contributors. International incidence of childhood cancer, 2001-10: a population-based registry study. Lancet Oncol. 2017 Jun;18(6):719-731. doi: 10.1016/S1470-2045(17)30186-9. Epub 2017 Apr 11. PMID 28410997
- [Background] Lam CG, Howard SC, Bouffet E, Pritchard-Jones K. Science and health for all children with cancer. Science. 2019 Mar 15;363(6432):1182-1186. doi: 10.1126/science.aaw4892. PMID 30872518
- [Background] Gohar SF, Comito M, Price J, Marchese V. Feasibility and parent satisfaction of a physical therapy intervention program for children with acute lymphoblastic leukemia in the first 6 months of medical treatment. Pediatr Blood Cancer. 2011 May;56(5):799-804. doi: 10.1002/pbc.22713. Epub 2011 Jan 16. PMID 21370414
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Katz ER, Seid M, Quiggins DJ, Friedman-Bender A, Castro CM. The Pediatric Cancer Quality of Life Inventory (PCQL). I. Instrument development, descriptive statistics, and cross-informant variance. J Behav Med. 1998 Apr;21(2):179-204. doi: 10.1023/a:1018779908502. PMID 9591169
- [Background] Varni JW, Burwinkle TM, Katz ER, Meeske K, Dickinson P. The PedsQL in pediatric cancer: reliability and validity of the Pediatric Quality of Life Inventory Generic Core Scales, Multidimensional Fatigue Scale, and Cancer Module. Cancer. 2002 Apr 1;94(7):2090-106. doi: 10.1002/cncr.10428. PMID 11932914
- [Background] Joffe L, Ladas EJ. Nutrition during childhood cancer treatment: current understanding and a path for future research. Lancet Child Adolesc Health. 2020 Jun;4(6):465-475. doi: 10.1016/S2352-4642(19)30407-9. Epub 2020 Feb 13. PMID 32061318
- [Background] Orgel E, Genkinger JM, Aggarwal D, Sung L, Nieder M, Ladas EJ. Association of body mass index and survival in pediatric leukemia: a meta-analysis. Am J Clin Nutr. 2016 Mar;103(3):808-17. doi: 10.3945/ajcn.115.124586. Epub 2016 Feb 10. PMID 26864366
- [Background] Ringwald-Smith K, Hill R, Evanoff L, Martin J, Sacks N. When Reality and Research Collide: Guidelines Are Essential for Optimal Nutrition Care in Pediatric Oncology. J Pediatr Hematol Oncol. 2022 Jan 1;44(1):e144-e151. doi: 10.1097/MPH.0000000000002200. PMID 34001795
- [Background] Fabozzi F, Trovato CM, Diamanti A, Mastronuzzi A, Zecca M, Tripodi SI, Masetti R, Leardini D, Muratore E, Barat V, Lezo A, De Lorenzo F, Caccialanza R, Pedrazzoli P. Management of Nutritional Needs in Pediatric Oncology: A Consensus Statement. Cancers (Basel). 2022 Jul 11;14(14):3378. doi: 10.3390/cancers14143378. PMID 35884438
- [Background] Tachibana H, Koga K, Fujimura Y, Yamada K. A receptor for green tea polyphenol EGCG. Nat Struct Mol Biol. 2004 Apr;11(4):380-1. doi: 10.1038/nsmb743. Epub 2004 Mar 14. PMID 15024383
- [Background] Garcia-Perdomo HA, Gomez-Ospina JC, Reis LO. Immunonutrition hope? Oral nutritional supplement on cancer treatment. Int J Clin Pract. 2021 Nov;75(11):e14625. doi: 10.1111/ijcp.14625. Epub 2021 Jul 19. PMID 34251725
- [Background] Palagyi A, Balane C, Shanthosh J, Jun M, Bhoo-Pathy N, Gadsden T, Canfell K, Jan S. Treatment abandonment in children with cancer: Does a sex difference exist? A systematic review and meta-analysis of evidence from low- and middle-income countries. Int J Cancer. 2021 Feb 15;148(4):895-904. doi: 10.1002/ijc.33279. Epub 2020 Sep 22. PMID 32875569
- [Background] Friedrich P, Lam CG, Itriago E, Perez R, Ribeiro RC, Arora RS. Magnitude of Treatment Abandonment in Childhood Cancer. PLoS One. 2015 Sep 30;10(9):e0135230. doi: 10.1371/journal.pone.0135230. eCollection 2015. PMID 26422208
- [Background] Gomez EV, Perez YM, Sanchez HV, Forment GR, Soler EA, Bertot LC, Garcia AY, del Rosario Abreu Vazquez M, Fabian LG. Antioxidant and immunomodulatory effects of Viusid in patients with chronic hepatitis C. World J Gastroenterol. 2010 Jun 7;16(21):2638-47. doi: 10.3748/wjg.v16.i21.2638. PMID 20518086
- [Background] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621
- [Background] Hernandez-Garcia S, Gonzalez V, Sanz E, Pandiella A. Effect of Oncoxin Oral Solution in HER2-Overexpressing Breast Cancer. Nutr Cancer. 2015;67(7):1159-69. doi: 10.1080/01635581.2015.1068819. Epub 2015 Aug 4. PMID 26241555
- [Background] Diaz-Rodriguez E, Hernandez-Garcia S, Sanz E, Pandiella A. Antitumoral effect of Ocoxin on acute myeloid leukemia. Oncotarget. 2016 Feb 2;7(5):6231-42. doi: 10.18632/oncotarget.6862. PMID 26756220
- [Background] Hernandez-Unzueta I, Benedicto A, Olaso E, Sanz E, Viera C, Arteta B, Marquez J. Ocoxin oral solution(R) as a complement to irinotecan chemotherapy in the metastatic progression of colorectal cancer to the liver. Oncol Lett. 2017 Jun;13(6):4002-4012. doi: 10.3892/ol.2017.6016. Epub 2017 Apr 10. PMID 28599406
- [Background] A teacupful of medicine? Nat Struct Mol Biol. 2008 Jun;15(6):537. doi: 10.1038/nsmb0608-537. PMID 18523460
- [Background] Siddiqui IA, Asim M, Hafeez BB, Adhami VM, Tarapore RS, Mukhtar H. Green tea polyphenol EGCG blunts androgen receptor function in prostate cancer. FASEB J. 2011 Apr;25(4):1198-207. doi: 10.1096/fj.10-167924. Epub 2010 Dec 21. PMID 21177307
- [Background] Milligan SA, Burke P, Coleman DT, Bigelow RL, Steffan JJ, Carroll JL, Williams BJ, Cardelli JA. The green tea polyphenol EGCG potentiates the antiproliferative activity of c-Met and epidermal growth factor receptor inhibitors in non-small cell lung cancer cells. Clin Cancer Res. 2009 Aug 1;15(15):4885-94. doi: 10.1158/1078-0432.CCR-09-0109. Epub 2009 Jul 28. PMID 19638461
- [Background] Yang C, Du W, Yang D. Inhibition of green tea polyphenol EGCG((-)-epigallocatechin-3-gallate) on the proliferation of gastric cancer cells by suppressing canonical wnt/beta-catenin signalling pathway. Int J Food Sci Nutr. 2016 Nov;67(7):818-27. doi: 10.1080/09637486.2016.1198892. Epub 2016 Jun 24. PMID 27338284
- [Background] Maruyama T, Murata S, Nakayama K, Sano N, Ogawa K, Nowatari T, Tamura T, Nozaki R, Fukunaga K, Ohkohchi N. (-)-Epigallocatechin-3-gallate suppresses liver metastasis of human colorectal cancer. Oncol Rep. 2014 Feb;31(2):625-33. doi: 10.3892/or.2013.2925. Epub 2013 Dec 13. PMID 24337301
- [Background] Roomi MW, Roomi N, Ivanov V, Kalinovsky T, Niedzwiecki A, Rath M. Inhibition of pulmonary metastasis of melanoma b16fo cells in C57BL/6 mice by a nutrient mixture consisting of ascorbic Acid, lysine, proline, arginine, and green tea extract. Exp Lung Res. 2006 Nov-Dec;32(10):517-30. doi: 10.1080/01902140601098552. PMID 17169857